CLINICAL TRIAL: NCT02292667
Title: Efficacy of the Ultrasound-guidedTransversus Abdominis Plane (TAP) Block on Postoperative Pain Control in Open Aortic Abdominal Aneurysm Repair Surgery
Brief Title: Efficacy of the Ultrasound-guided Transversus Abdominis Plane Block in Open Aortic Abdominal Aneurysm Repair Surgery
Acronym: ETAP
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire de Besancon (Other)
Responsible Party: Principal Investigator, Julien CHENET, M.D., Centre Hospitalier Universitaire de Besancon
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: API/2014/52; 2014-003665-20 (EudraCT Number)
Record Dates: First submitted 2014-11-05; First posted 2014-11-17 (Estimated); Last update posted 2016-08-12 (Estimated); Status verified 2016-08

CONDITIONS: Aortic Aneurysm, Abdominal; Pain; Anesthesia, Local
Keywords: Transversus Abdominis Plane Block; Postoperative Pain Management; Open Repair of Aortic Abdominal Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Pain | interventions — Passive Cutaneous Anaphylaxis; Analgesia, Patient-Controlled; Acetaminophen

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TAP BLOCK (Experimental): Patients included in the ETAP group will receive the combination of a bilateral ultrasound-guided Transversus Abdominis Plane (TAP) block and a multimodal intravenous analgesia protocol for the postoperative pain management after the surgical open repair of an aortic abdominal aneurysm.
  The TAP block consists in 2 ultrasound-guided injections of Ropivacaine 0.375% on each side of the abdominal wall between the internal oblique and transversus abdominis muscles: 1 subcostal injection and 1 supra-iliac injection (i.e 10 ml of Ropivacaine 0.375% by injection).
  The multimodal intravenous analgesia protocol consists in the association of intravenous infusion of 1 g of Acetaminophen every 6 h and intravenous patient-controlled analgesia (PCA) with Chlorhydrate of Morphine 1 mg/ml.
  Interventions: Procedure: TAP block; Drug: PCA with Chlorhydrate of Morphine; Drug: Acetaminophen
- CONTROL (Active Comparator): Patients included in the CONTROL group will receive a multimodal intravenous analgesia protocol alone for the postoperative pain management after the surgical open repair of an aortic abdominal aneurysm.
  The multimodal intravenous analgesia protocol consists in the association of intravenous infusion of 1 g of Acetaminophen every 6 h and intravenous patient-controlled analgesia (PCA) with Chlorhydrate of Morphine 1 mg/ml.
  Interventions: Drug: PCA with Chlorhydrate of Morphine; Drug: Acetaminophen

INTERVENTIONS:
Procedure: TAP block — The aim of the Transversus Abdominis Plane (TAP) Block is to deposit local anesthetic in the plane between the internal oblique and the transversus abdominis muscles targeting the spinal nerves in this plane. The local anesthetic used in the ETAP study is Ropivacaine 0.375%. 2 ultrasound-guided injections of 10 ml will be performed on each side of the abdominal wall: 1 subcostal injection and 1 supra-iliac injection.
  Other Names: Transversus Abdominis Plane Block
  Arms: TAP BLOCK
Drug: PCA with Chlorhydrate of Morphine — Doses of 1 mg of Chlorhydrate of Morphine will be delivered intravenously by the Patient Controlled Analgesia (PCA) pump. The PCA pump is a computerized pump which contains a syringe of 1 mg/ml of Chlorhydrate of Morphine as prescribed by the physician in charge of the patient, and connected directly to a patient's intravenous line. Doses of Chlorhydrate of Morphine can be self-administered by the patient as needed by the having the patient press a button.
  Other Names: Patient Controlled Analgesia (PCA)
Drug: Acetaminophen — 1 g of Acetaminophen will be given intravenously each 6 h during 48 hours after the surgical procedure.
  Other Names: Paracetamol

SUMMARY:
The ETAP study aim to assess the effect of the addition of an ultrasound-guided transversus abdominis plane (TAP) block to a multimodal intravenous analgesia protocol on the postoperative pain control in open surgical repair of abdominal aortic aneurysm. The ETAP study is a single-center open-label randomized controlled trial. Half of patients included will receive the association of TAP block and multimodal intravenous analgesia, and the other half will receive the multimodal intravenous analgesia alone. The multimodal intravenous analgesia includes intravenous paracetamol and intravenous patient-controlled analgesia with morphine.

DETAILED DESCRIPTION:
The open repair of abdominal aortic aneurysm (AAA) is a painful surgery. Patients suffering from AAA are at high risk of perioperative cardiovascular and pulmonary complications. It has been previously suggested that a bad perioperative pain control could increase the incidence of such complications.

Intravenous patient-controlled analgesia (PCA) with morphine is widely considered as the gold standard treatment of the postoperative pain in open repair of AAA. High dose of morphine are often required and could delay the postoperative recovery and discharge. Side effects of morphine, such as respiratory depression, nausea, vomiting or pruritus, are responsible for patient discomfort and dissatisfaction when high doses are used.

The efficacy of the ultrasound-guided transversus abdominis plane (TAP) block has been described for pain management following abdominal surgery, such as gastrectomy or kidney transplantation. The efficacy of the association of TAP block and PCA with morphine was higher than multimodal intravenous analgesia including PCA with morphine and than the combination of PCA with morphine and epidural analgesia. To our knowledge, the efficacy of the ultrasound-guided TAP block has never been studied for the postoperative pain control in AAA surgery.

ELIGIBILITY:
Inclusion Criteria:

* ASA (American Society of Anesthesiologists) physical status 1, 2 or 3
* Elective surgery for open repair of an aortic abdominal aneurysm performed in the Vascular Surgery Unit of the University Hospital of Besancon
* Informed consent given
* Health medical insurance affiliation

Exclusion Criteria:

* Poor adherence to protocol attended
* Incapacity to consent
* Pregnancy and/or breast feeding
* Endovascular repair of aortic abdominal aneurysm
* Emergent surgery of a rupture or a fissuration of aortic abdominal aneurysm
* Chronic medical treatment by clopidogrel if clopidogrel not stopped 5 days before surgery at least
* Chronic medical treatment by prasugrel if prasugrel not stopped 7 days before surgery at least
* Chronic medical treatment by ticlopidine, inhibitors of phosphodiesterase , inhibitors of glycoprotein IIb/IIIa, adenosine triphosphate analogs or thrombin receptor antagonists
* Congenital or acquired bleeding disorder
* Incapacity to use patient-controlled analgesia device
* Chronic opioid abuse or dependence
* Chronic renal failure defined as a clearance < 30 ml/min
* Severe hepatic failure
* Other contraindications to ropivacaïne (allergy, medical history of porphyria, hypovolemia)
* Contraindications to acetaminophen
* Contraindications to morphine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-01; Primary Completion 2018-12 (Estimated); Study Completion 2019-01 (Estimated)

PRIMARY OUTCOMES:
Morphine consumption during the first postoperative 24 hours | 24 hours
  The morphine consumption during the first postoperative 24 hours is the total dose of morphine delivered both by the patient-controlled analgesia device and during the titration of morphine by the nurse in the post-anesthesia care unit.

SECONDARY OUTCOMES:
Delay between the last peroperative injection of opioid and the first administration of morphine in the post-anesthesia care unit | 24 hours
Morphine consumption during the first postoperative 48 hours | 48 hours
  The morphine consumption during the first postoperative 48 hours is the total dose of morphine delivered both by the patient-controlled analgesia device and during the titration of morphine by the nurse in the post-anesthesia care unit.
Pain intensity at rest assessed by the visual analog scale for pain | 48 hours
Pain intensity at mobilisation assessed by the visual analog scale for pain | 48 hours
Percentage of patients suffering from insomnia during the first and/or the second postoperative night | 48 hours
Percentage of patients suffering from awakenings during the first and/or the second postoperative night | 48 hours
Incidence of morphine side effects | 48 hours
  Morphine side effects include: nausea, vomiting, pruritus, drowsiness, respiratory depression
Incidence of TAP block side effects | 48 hours
  TAP block side effects are any side effect occuring in the ETAP group and considered to be related to the TAP block by the safety board of the study.
Ropivacaine sides effects | 48 hours
  Ropivacaine sides effects are: cardiac toxicity, neurologic toxicity, allergy
Post-operative morbidity | Day 30
  Any of the following events occuring within the 30 first post-operative days: myocardial infarction, acute congestive heart failure, ventricular tachycardia, ventricular fibrillation, atelectasis, pneumonia, acute respiratory failure requiring invasive or non invasive mechanical ventilation, acute kidney failure, non infectious systemic inflammatory response syndrome, sepsis, surgical wound complication.
30-day survival | Day 30
Duration of hospital stay | Expected average of 10 days
  Patients will be followed for the duration of hospital stay, an expected average of 10 days.

CONTACTS AND LOCATIONS:
Overall Officials: Julien Chenet, MD, Principal Investigator — Centre Hospitalier Régional Universitaire de Besancon
Locations (1):
- CHU Besançon, Besançon, Doubs, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] McDonnell JG, Curley G, Carney J, Benton A, Costello J, Maharaj CH, Laffey JG. The analgesic efficacy of transversus abdominis plane block after cesarean delivery: a randomized controlled trial. Anesth Analg. 2008 Jan;106(1):186-91, table of contents. doi: 10.1213/01.ane.0000290294.64090.f3. PMID 18165577